CLINICAL TRIAL: NCT03269630
Title: New Orleans Pulmonary Hypertension Biobank
Acronym: NO-PH Biobank
Status: Recruiting | Type: Observational
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Matthew Lammi, Associate Professor of Medicine, Louisiana State University Health Sciences Center in New Orleans
Other Study IDs: LSU
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Hypertension; Systemic Sclerosis; Mixed Connective Tissue Disease; Heart Failure With Normal Ejection Fraction; Healthy
MeSH Terms: conditions — Hypertension, Pulmonary; Scleroderma, Systemic; Mixed Connective Tissue Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (serum, plasma, buffy coat, PBMCs) Urine Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Clinic patients (Comprehensive Pulmonary Hypertension Center): * Pulmonary hypertension patients (WHO group 1-5)
  * Systemic sclerosis patients without pulmonary hypertension
  * Mixed connective tissue disease patients without pulmonary hypertension
  Interventions: Other: No intervention. Biospecimen collection only
- Outpatient right heart catheterization patients: -Outpatients undergoing right heart catheterization for any indication
  Interventions: Other: No intervention. Biospecimen collection only
- Healthy controls: * Age>18
  * Not actively smoking
  * No chronic medical conditions
  Interventions: Other: No intervention. Biospecimen collection only

INTERVENTIONS:
Other: No intervention. Biospecimen collection only — Biospecimen collection

SUMMARY:
Pulmonary hypertension (PH) is a serious condition characterized by a mean pulmonary artery pressure >=25mmHg on right heart catheterization (RHC). Despite advances in PH care, outcomes are still sub-optimal and further research is required into the pathobiology of the disease and development of biomarkers that can guide clinical care. The investigators are establishing a biobank to collect samples (blood, urine, stool) from patients with pulmonary hypertension, patients at high risk for pulmonary hypertension, healthy controls, and patients undergoing right heart catheterization. Specimens will be stored for future investigations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pulmonary hypertension and followed at the Comprehensive Pulmonary Hypertension Center OR
* Diagnosis of systemic sclerosis and followed at the Comprehensive Pulmonary Hypertension Center OR
* Diagnosis of mixed connective tissue disease and followed at the Comprehensive Pulmonary Hypertension Center OR
* Undergoing outpatient right heart catheterization

Exclusion Criteria:

* Age<18
* Pregnant
* Unable to understand English
* Currently incarcerated
* Unwilling or unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled from 2 venues: 1) Comprehensive Pulmonary Hypertension Center clinic (pulmonary hypertension, systemic sclerosis without PH, mixed connective tissue disease without PH) and 2) Outpatient right heart catheterization lab. Healthy subjects (age>18, not currently smoking, no chronic medical conditions) will also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2017-12-29 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Collection of biospecimens | 10 years
  Biospecimen collection only

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center-New Orleans, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A sharing plan will be developed to share biospecimens with interested researchers.